CLINICAL TRIAL: NCT00409487
Title: Comparative Study of Effect of Valsartan 160mg Treatment Versus Continuous Positive Airway Pressure on Arterial Blood Pressure in Patients Who Have an Obstructive Sleep Apnea Syndrome and a Weak or Moderate Hypertension.
Brief Title: Effects of Continuous Positive Airway Pressure and Valsartan Treatments on Arterial Blood Pressure in OSAS Patients
Acronym: VALSAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: University Hospital, Grenoble, Délégation de la Recherche Clinique et de l'Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0617
Record Dates: First submitted 2006-12-08; First posted 2006-12-11 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Hypertension,; Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; hypertension; ambulatory bloop pressure monitoring
MeSH Terms: conditions — Hypertension; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 8 weeks of Valsartant treatment, 4 weeks of washout, 8 weeks of CPAP and 8 weeks of Valsartant plus CPAP treatments
  Interventions: Device: Continuous positive airway pressure (CPAP); Drug: Valsartant treatment
- 2 (Experimental): 8 weeks of CPAP , 4 weeks of washout, 8 weeks of Valsartant treatment and 8 weeks of Valsartant plus CPAP treatments
  Interventions: Device: Continuous positive airway pressure (CPAP); Drug: Valsartant treatment

INTERVENTIONS:
Device: Continuous positive airway pressure (CPAP) — 8 weeks of CPAP
  Other Names: CPAP treatment
Drug: Valsartant treatment — 8 weeks of Valsartant treatment (160 mg / day)

SUMMARY:
The main objective of the study is to compare the decrease of mean arterial blood pressure over 24 hours in patients having obstructive sleep apnea syndrome and weak or moderate hypertension, treated by Valsartan 160mg per day versus continuous Positive Airway Pressure.

DETAILED DESCRIPTION:
It is now well known that cardiovascular risks are increased in patients with obstructive sleep apnea syndrome (OSAS). Also a link has already been demonstrated between OSAS and hypertension.

Nowadays, the most efficient treatment of the OSAS is the continuous Positive Airway Pressure (cPAP). Several studies have also shown that cPAP could reduce arterial blood pressure of about 3,3 mmHg in OSAS patients. Unfortunately, 40% of the patients either refuse being treated by cPAP or give up treatment. In parallel, alternative medications are proposed to patients with moderate OSAS and hypertension, in order to decrease their cardiovascular risks. A study led on rats has shown the superiority of the beta adrenergic blocking agents in the decrease of hypertension in OSAS patients.

Our study has also the objective to compare the effects of Valsartan and cPAP on hypertension in OSAS patients. Those one will be randomized either in the group "treatment by Valsartan and then by cPAP" or in the group "treatment by cPAP and then Valsartan" (cross-over study).

ELIGIBILITY:
Inclusion Criteria:

* male/female over than 18 years old
* patient with an obstructive sleep apnea (apnea-hypopnea index > or equal to 15)
* patient with weak or moderate hypertension (140 <= SBP < 180 mmHg and 90 <= DBP < 110 mmHg). Patient with antihypertensive monotherapy must stop their treatment and respect a washout period of at least 4 weeks before the screening visit. For patient treated by antialdosterone, the washout period will be of at least 8 weeks.
* negative pregnancy test
* ambulatory patient
* patient who have signed the informed consent form
* patient affiliated to social security

Exclusion Criteria:

* pregnant or nursing woman
* woman who refuses to use contraceptive method
* acute hepatic failure, biliary cirrhosis, cholestasis
* clearance of Cockcroft < 30 ml/min/1.73m2
* kaliemia >= 5.5 mmol/l
* acute hypertension (SBP>= 180 mmHg and/or DBP >= 110 mmHg)
* acute daytime sleepiness (Epworth rating scale > 15)
* patient with a profession that is inconsistent with the continuous positive airway pressure (CPAP) treatment
* known cardiovascular pathologies
* contraindication to CPAP
* allergy to Valsartan
* patient treated with lithium
* patient treated with drug(s) acting on arterial blood pressure
* patient on tutelle or curatelle
* patient kept in detention, major protected by the law, hospitalised person
* patient currently participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-12; Primary Completion 2006-12 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
ambulatory blood pressure monitoring over 24 hours, at inclusion visit (day=0), 8 weeks, 12 weeks, and 20 weeks | 24 h

SECONDARY OUTCOMES:
clinical blood pressure measurement at inclusion, 8 weeks, 12 weeks, and 20 weeks; pulse wave speed at inclusion, 8 weeks, 12 weeks, and 20 weeks; baroreceptor reflex at inclusion, 8 weeks, 12 weeks, and 20 weeks. | 1 h

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis JL PEPIN, ProfessorPhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, Grenoble, France

REFERENCES:
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; National Heart, Lung, and Blood Institute Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure; National High Blood Pressure Education Program Coordinating Committee. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure: the JNC 7 report. JAMA. 2003 May 21;289(19):2560-72. doi: 10.1001/jama.289.19.2560. Epub 2003 May 14. PMID 12748199
- [Background] Baguet JP, Hammer L, Levy P, Pierre H, Rossini E, Mouret S, Ormezzano O, Mallion JM, Pepin JL. Night-time and diastolic hypertension are common and underestimated conditions in newly diagnosed apnoeic patients. J Hypertens. 2005 Mar;23(3):521-7. doi: 10.1097/01.hjh.0000160207.58781.4e. PMID 15716692
- [Background] Baguet JP, Narkiewicz K, Mallion JM. Update on Hypertension Management: obstructive sleep apnea and hypertension. J Hypertens. 2006 Jan;24(1):205-8. doi: 10.1097/01.hjh.0000198039.39504.63. No abstract available. PMID 16331122
- [Background] Pepperell JC, Ramdassingh-Dow S, Crosthwaite N, Mullins R, Jenkinson C, Stradling JR, Davies RJ. Ambulatory blood pressure after therapeutic and subtherapeutic nasal continuous positive airway pressure for obstructive sleep apnoea: a randomised parallel trial. Lancet. 2002 Jan 19;359(9302):204-10. doi: 10.1016/S0140-6736(02)07445-7. PMID 11812555
- [Background] Becker HF, Jerrentrup A, Ploch T, Grote L, Penzel T, Sullivan CE, Peter JH. Effect of nasal continuous positive airway pressure treatment on blood pressure in patients with obstructive sleep apnea. Circulation. 2003 Jan 7;107(1):68-73. doi: 10.1161/01.cir.0000042706.47107.7a. PMID 12515745
- [Background] Kraiczi H, Hedner J, Peker Y, Grote L. Comparison of atenolol, amlodipine, enalapril, hydrochlorothiazide, and losartan for antihypertensive treatment in patients with obstructive sleep apnea. Am J Respir Crit Care Med. 2000 May;161(5):1423-8. doi: 10.1164/ajrccm.161.5.9909024. PMID 10806134
- [Background] Jordan J, Engeli S, Boschmann M, Weidinger G, Luft FC, Sharma AM, Kreuzberg U. Hemodynamic and metabolic responses to valsartan and atenolol in obese hypertensive patients. J Hypertens. 2005 Dec;23(12):2313-8. doi: 10.1097/01.hjh.0000188734.98463.82. PMID 16269974
- [Background] Calvo C, Hermida RC, Ayala DE, Ruilope LM. Effects of telmisartan 80 mg and valsartan 160 mg on ambulatory blood pressure in patients with essential hypertension. J Hypertens. 2004 Apr;22(4):837-46. doi: 10.1097/00004872-200404000-00028. PMID 15126927
- [Background] Baguet JP, Pepin JL, Hammer L, Levy P, Mallion JM. [Cardiovascular consequences of obstructive sleep apnea syndrome]. Rev Med Interne. 2003 Aug;24(8):530-7. doi: 10.1016/s0248-8663(03)00142-5. French. PMID 12888174
- [Derived] Pepin JL, Tamisier R, Barone-Rochette G, Launois SH, Levy P, Baguet JP. Comparison of continuous positive airway pressure and valsartan in hypertensive patients with sleep apnea. Am J Respir Crit Care Med. 2010 Oct 1;182(7):954-60. doi: 10.1164/rccm.200912-1803OC. Epub 2010 Jun 3. PMID 20522795